CLINICAL TRIAL: NCT03485222
Title: EMPA-TROPISM Trial: Are the "Cardiac Benefits" of Empagliflozin Independent of Its Hypoglycemic Activity?
Brief Title: Are the "Cardiac Benefits" of Empagliflozin Independent of Its Hypoglycemic Activity? (ATRU-4).
Acronym: EMPA-TROPISM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Boehringer Ingelheim (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Juan Badimon, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 17-2457
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Results first posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular diseases; Heart Failure; LV remodeling; SGLT-2 Inhibitors; Empagliflozin; Cardiac MRI
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Experimental): 10mg once a day
  Interventions: Drug: Empagliflozin
- Placebos (Placebo Comparator): placebo once a day
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Empagliflozin — 6 months
  Arms: Empagliflozin
Drug: Placebos — placebo equivalent for 6 months
  Arms: Placebos

SUMMARY:
Purpose:

The overall hypothesis of the study is that the benefits attained in the EMPA-OUTCOME were, at least in part, mediated by a glucose-independent mechanism. Thus, to demonstrate the existence of the postulated non-glucose dependent effects, the researchers will investigate the safety and efficacy of empagliflozin versus placebo on top of guideline-directed medical therapy in heart failure patients with reduced ejection fraction without diabetes.

DETAILED DESCRIPTION:
Heart failure (HF) is a frequent co-morbid condition associated with poor prognosis in diabetes, particularly among older patients. HF accounts for more than 1 Million hospitalizations annually in USA. In addition, HF hospitalizations are associated with significant high risk of post-discharge mortality and recurrent hospitalizations. Almost one-half of patients will be re-hospitalized within 6 months and one-third will die within 12 months of discharge. Median survival after HF diagnosis is about 5 years and is similar for HFpEF and heart failure with reduced ejection fraction (HFrEF) patients. Diabetes as co-morbidity multiplies risk of hospital admissions in HF patients.

Type 2 Diabetes Mellitus (T2DM) is a pathological condition characterized by elevated glucose levels and it is associated with high incidence of cardiovascular (CV) events. Several hypoglycemic agents have successfully managed the elevated glucose levels but with little or no impact on CV events. Management of concomitant HF in T2DM is particularly challenging, as some glucose-lowering agents, such as TZDs, are contraindicated in the treatment of HF patients. Thus, there was a need for an oral agent that improved glycemia as well as provided CV benefits. Empagliflozin is the first glucose-lowering agent showing that not only improves glycemic control but also has cardiovascular benefits. The recent EMPA-OUTCOME trial has shown significant reductions in major adverse cardiac events (MACE), cardiovascular mortality, and hospitalization for Heart Failure (HF) by Empagliflozin given on top of standard-of-care therapy for T2DM patients with Cardiovascular disease (CVD). The dramatic change driving the superiority of the primary composite outcome was a significantly lower CV death rate (38% relative risk reduction). In addition, there were also an impressive 35% and 38% relative risk reductions in hospitalization for heart failure (HF) and death from any cause, respectively.

Empagliflozin is a member of a new class of hypoglycemic agents, the SGLT-2 inhibitors. There are a couple of characteristics that single out the SGLT2 inhibitors from other hypoglycemic drugs. One is their low hypoglycemic risk since they act on the urinary excretion of glucose without interfering with the physiologic response to hypoglycemia. And the other is their "positive" cardiovascular effects such as lowering blood pressure, arterial stiffness, urinary microalbuminuria and triglycerides while increasing HDL-Cholesterol levels. Therefore, the combination of the above-mentioned observations led to some investigators to suggest that these benefits may be, at least in part, independent of its hypoglycemic activity and thus, Empagliflozin could be considered a "cardiac" drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients should meet the following inclusion criteria:
* Ambulatory patients age 18-85 years
* Diagnosis of Heart failure (NYHA II to III)
* LVEF<50% on echocardiography or CMRI in the previous 6 months
* Have stable symptoms and therapy for HF within the last 3 months.

Exclusion Criteria:

* Pregnant or lactating women.
* Any history of diabetes by medical history or by any of the established criteria by the American Diabetes Association. It also includes patients with history of diabetes in remission.
* ACS or cardiac surgery within the last 3 months.
* Cancer or any other life-threatening condition.
* Pancreatitis.
* Glomerular Filtration Rate < 45 ml/Kg/min.
* Use of continuous parental inotropic agents.
* Systolic BP < 90 mm Hg.
* Psychiatric disease incompatible with being in study.
* Any contraindication to MRI procedures.
* Any other medical or physical condition considered to be inappropriate by a study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Badimon, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Heart - Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Santos-Gallego CG, Vargas-Delgado AP, Requena-Ibanez JA, Garcia-Ropero A, Mancini D, Pinney S, Macaluso F, Sartori S, Roque M, Sabatel-Perez F, Rodriguez-Cordero A, Zafar MU, Fergus I, Atallah-Lajam F, Contreras JP, Varley C, Moreno PR, Abascal VM, Lala A, Tamler R, Sanz J, Fuster V, Badimon JJ; EMPA-TROPISM (ATRU-4) Investigators. Randomized Trial of Empagliflozin in Nondiabetic Patients With Heart Failure and Reduced Ejection Fraction. J Am Coll Cardiol. 2021 Jan 26;77(3):243-255. doi: 10.1016/j.jacc.2020.11.008. Epub 2020 Nov 13. PMID 33197559
- [Derived] Angermann CE, Sehner S, Gerhardt LMS, Santos-Gallego CG, Requena-Ibanez JA, Zeller T, Maack C, Sanz J, Frantz S, Ertl G, Badimon JJ. Anaemia predicts iron homoeostasis dysregulation and modulates the response to empagliflozin in heart failure with reduced ejection fraction: the EMPATROPISM-FE trial. Eur Heart J. 2025 Apr 22;46(16):1507-1523. doi: 10.1093/eurheartj/ehae917. PMID 39907687
- [Derived] Angermann CE, Santos-Gallego CG, Requena-Ibanez JA, Sehner S, Zeller T, Gerhardt LMS, Maack C, Sanz J, Frantz S, Fuster V, Ertl G, Badimon JJ. Empagliflozin effects on iron metabolism as a possible mechanism for improved clinical outcomes in non-diabetic patients with systolic heart failure. Nat Cardiovasc Res. 2023 Nov;2(11):1032-1043. doi: 10.1038/s44161-023-00352-5. Epub 2023 Oct 26. PMID 39196095
- [Derived] Kanie T, Mizuno A, Takaoka Y, Suzuki T, Yoneoka D, Nishikawa Y, Tam WWS, Morze J, Rynkiewicz A, Xin Y, Wu O, Providencia R, Kwong JS. Dipeptidyl peptidase-4 inhibitors, glucagon-like peptide 1 receptor agonists and sodium-glucose co-transporter-2 inhibitors for people with cardiovascular disease: a network meta-analysis. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD013650. doi: 10.1002/14651858.CD013650.pub2. PMID 34693515
- [Derived] Requena-Ibanez JA, Santos-Gallego CG, Rodriguez-Cordero A, Vargas-Delgado AP, Mancini D, Sartori S, Atallah-Lajam F, Giannarelli C, Macaluso F, Lala A, Sanz J, Fuster V, Badimon JJ. Mechanistic Insights of Empagliflozin in Nondiabetic Patients With HFrEF: From the EMPA-TROPISM Study. JACC Heart Fail. 2021 Aug;9(8):578-589. doi: 10.1016/j.jchf.2021.04.014. PMID 34325888

RESULTS

PARTICIPANT FLOW:
Groups:
- Empagliflozin: 10mg once a day for 6 months
- Placebos: Placebo equivalent once a day for 6 months
Period: Overall Study
Arm/Group | Empagliflozin | Placebos
Started | 42 | 42
Completed | 40 | 40
Not Completed | 2 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin | Placebos | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (10.9) | 59.9 (13.1) | 62 (12.1)
Age, Customized [Count of Participants; unit: Participants]
  <65 yrs | 24 | 28 | 52
  >65 yrs | 18 | 14 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 27 | 27 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 7 | 23
  Hispanic/Latino | 19 | 23 | 42
  African American | 7 | 9 | 16
  Asian | 0 | 3 | 3
Hypertension [Count of Participants; unit: Participants] | 34 | 28 | 62
Hyperlipidemia [Count of Participants; unit: Participants] | 32 | 30 | 62
Cigarette smoking (past or present) [Count of Participants; unit: Participants] | 18 | 12 | 30
Atrial fibrillation [Count of Participants; unit: Participants] | 10 | 8 | 18
Cause of Heart Failure (HF) [Count of Participants; unit: Participants]
  Ischemic | 23 | 19 | 42
  Nonischemic | 19 | 23 | 42
Devices [Count of Participants; unit: Participants] — Implantable cardioverter-defibrillator (ICD), Cardiac resynchronization therapy (CRT), Pacemaker
  Participants | 9 | 8 | 17
Statin History [Count of Participants; unit: Participants] | 33 | 30 | 63
Number of participants taking ACE inhibitor/ARB (alone) at baseline [Count of Participants; unit: Participants] | 16 | 19 | 35
Angiotensin receptor-neprilysin inhibitor (ARNi) [Count of Participants; unit: Participants] | 21 | 15 | 36
B-blockers [Count of Participants; unit: Participants] | 36 | 38 | 74
Loop diuretics [Count of Participants; unit: Participants] | 22 | 24 | 46
Thiazide diuretics [Count of Participants; unit: Participants] | 3 | 2 | 5
Mineralocorticoid antagonists [Count of Participants; unit: Participants] | 13 | 15 | 28
Ca-blockers [Count of Participants; unit: Participants] | 5 | 5 | 10
Antiplatelet [Count of Participants; unit: Participants] | 29 | 26 | 55
Anticoagulants [Count of Participants; unit: Participants] | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricle-end Systolic Volume (ESV)
Description: End-systolic volume (ESV) is the volume of blood in a ventricle at the end of contraction of the left ventricle (LV). Change from baseline to study end at 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Empagliflozin | Placebos
Number analyzed (Participants) | 40 | 40
ml | -26.6 (20.5) | -0.5 (21.9)

2. Primary Outcome: Change in LV-end Diastolic Volume (EDV)
Description: End-diastolic volume (EDV) is the volume of blood in the left ventricle at end load or filling in (diastole) or the amount of blood in the ventricles just before systole. Change from baseline to study end at 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Empagliflozin | Placebos
Number analyzed (Participants) | 40 | 40
ml | -25.1 (26) | -1.5 (25.4)

3. Secondary Outcome: Change in LV-Ejection Fraction Index
Description: The volumetric fraction of blood ejected from the left ventricle of the heart with each heartbeat. Change from baseline to study end at 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: percent ejection fraction
Arm/Group | Empagliflozin | Placebos
Number analyzed (Participants) | 40 | 40
percent ejection fraction | 6.0 (4.2) | -0.1 (3.9)

4. Secondary Outcome: Change in VO2 Consumption
Description: Oxygen consumption - the amount of oxygen consumed by the tissues of the body, usually measured as the oxygen uptake in the lung, also called the V02max measure. Change from baseline to study end at 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | Empagliflozin | Placebos
Number analyzed (Participants) | 40 | 40
ml/min/kg | 1.1 (2.6) | -0.5 (1.9)

5. Secondary Outcome: Change in 6 Min Walk Test
Description: The distance covered over a time of 6 minutes. Change from baseline to study end at 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Empagliflozin | Placebos
Number analyzed (Participants) | 40 | 40
m | 81 (64) | -35 (68)

6. Secondary Outcome: Change in Kansas Cardiomyopathy Questionnaire (KCCQ-12)
Description: The KCCQ-12 is an instrument most widely used to evaluate QoL in Heart Failure (HF) patients. It is a questionnaire containing 12 questions with full scores ranging from 12 (poor quality of life) to 70 (good quality of life). Higher score indicates better quality of life. Change from baseline to study end at 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empagliflozin | Placebos
Number analyzed (Participants) | 40 | 40
score on a scale | 21 (18) | 1.9 (15)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Empagliflozin | Placebos
All-Cause Mortality (participants affected / at risk) | 0/40 | 1/40
Serious Adverse Events (participants affected / at risk) | 1/40 | 2/40
Other Adverse Events (participants affected / at risk) | 2/40 | 1/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin (N=40) | Placebos (N=40)
Malignant Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Worsening Heart Failure (Cardiac disorders) | 0 | 1
New ICD Implant (Cardiac disorders) | 1 | 2
New Cardiomems Implant (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin (N=40) | Placebos (N=40)
Hepatic Injury (Hepatobiliary disorders) | 0 | 1 — ALT and/or AST ≥ 5 fold ULN
Migraine (Nervous system disorders) | 1 | 0
Motor Vehicle Accident (Social circumstances) | 1 | 0

LIMITATIONS AND CAVEATS:
This is a single-site trial with a relatively small number of patients; however, the high reproducibility of CMR allows for the utilization of reduced sample sizes. A second limitation is the relatively high number of dropouts in the CPET. Third, this trial have exclusively studied heart failure with reduced ejection fraction(HFrEF) patients; whether patients with heart failure with preserved ejection fraction can benefit from SGLT2i cannot be answered by this study and remains to be determined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT03485222/Prot_SAP_001.pdf